CLINICAL TRIAL: NCT05951465
Title: Determination of the Median Effective Dose of Propofol in Combination With Different Doses of Esketamine During Colonoscopy for Children With Autism Spectrum Disorder
Brief Title: Esketamine and Propofol for Children With Autism Spectrum Disorder Undergoing Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Collaborators: Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: esketamine 2023 N002
Record Dates: First submitted 2023-05-25; First posted 2023-07-19 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-05

CONDITIONS: Autism Spectrum Disorder
Keywords: colonoscopy; anaesthesia; autism spectrum disorder; propofol; esketamine
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Esketamine; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eskatemine 0.3mg/kg + propofol (Experimental): eskatemine dose will be 0.3 mg/kg. Propofol dose for the first patient will be 2.5mg/kg. Doses for the subsequent patients will increase or decrease by 0.8 mg/kg using the Dixon Up and Down method.
  Interventions: Drug: Esketamine; Drug: Propofol
- eskatemine 0.6mg/kg + propofol (Experimental): eskatemine dose will be 0.6 mg/kg. Propofol dose for the first patient will be 2.0mg/kg. Doses for the subsequent patients will increase or decrease by 0.4 mg/kg using the Dixon Up and Down method.
  Interventions: Drug: Esketamine; Drug: Propofol

INTERVENTIONS:
Drug: Esketamine — esketamine dose will be 0.3 mg/kg. Propofol dose for the first patient will be 2.5 mg/kg. Doses for the subsequent patients will increase or decrease by 0.8 mg/kg using the Dixon Up and Down method.
  Arms: eskatemine 0.3mg/kg + propofol
Drug: Esketamine — esketamine dose will be 0.6 mg/kg. Propofol dose for the first patient will be 2.0 mg/kg. Doses for the subsequent patients will increase or decrease by 0.4 mg/kg using the Dixon Up and Down method.
  Arms: eskatemine 0.6mg/kg + propofol
Drug: Propofol — propofol

SUMMARY:
The purpose of this study is to examine the dose-response relationship of esketamine in combination with propofol for children with Autism Spectrum Disorder undering colonoscopy.

DETAILED DESCRIPTION:
Autistic children appear with significant frequency for medical services, lots of which requiring procedural sedation or anaesthesia. They have often been described as difficult to sedate or anesthetize due to a variety of ASD symptoms. It is a challenging task to provide safe and effective sedation during the colonoscopic procedure in autism children. Propofol sedation for endoscopic procedures is safe and acceptable for children, especially those who express significant anxiety. Propofol-based sedation turned out to be the most effective dosage regimens, with effectiveness comparable to general anesthesia. The addition of certain dose ketamine to propofol may increase the effectiveness without creating more adverse events.

ELIGIBILITY:
Inclusion Criteria:

* （1) aged 2-12 years;
* (2) diagnosed with ASD by pediatric psychiatrists in accordance with the criteria in the Fifth Edition of Diagnostic and Statistical Manual of Mental Disorders (DSM-V);
* (3) evaluated as American Society of Anesthesiologists (ASA) physical status I-II;
* (4) scheduled for colonic procedure.

Exclusion Criteria:

* (1) oral sedation (premedication) before intravenous catheter placement;
* (2) any contraindication to study medications;
* (3) other circumstances in which the investigator determined that a patient was not suitable for participation in the clinical trial.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Dose of Propofol Required to Prevent Movement (Response) to Insertion of colonoscpopy 1 | Procedure (This outcome is measured at the time of insertion of colonoscopy)
  The objective is to determine the effective bolus dose in 50% of subjects (ED50) of propofol in combination with ketamine 0.3, 0.6mg/kg that produces an adequate depth of anesthesia to prevent minimal or no movement on colonoscopy insertion in children with Autism spectrum disorder.
Dose of Propofol Required to Prevent Movement (Response) to Insertion of colonoscpopy 2 | Procedure (This outcome is measured at the time of insertion of colonoscopy)
  The objective is to determine the effective bolus dose in 95% of subjects (ED50) of propofol in combination with ketamine 0.3, 0.6mg/kg that produces an adequate depth of anesthesia to prevent minimal or no movement on colonoscopy insertion in children with Autism spectrum disorder.

SECONDARY OUTCOMES:
movement score during the procedure | during the procudure
  (1 = no movement; 2 = semipurposeful allowing continuation of the procedure; 3 = vigorous purposeful movements withholding the procedure)
arterial blood pressure | during the procudure
  arterial blood pressure was measured noninvasively at four time points:T0: before induction of sedation,T1: immediately after induction of sedation, T2: complete evaluation of the coln through colonoscopy, T3: at the end of colonic TET procedure。
adverse event | during the procedure - 24 hours after procedure
  (including hypoxia (SpO2 <93% for >10 s) or respiratory depression (apnea >15 s), hypotension (MAP < 20% from baseline) or bradycardia (HR < 60 x/min and/or decrease in HR > 20% from baseline) were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Hospital, Nanjing, Jiangsu, China